CLINICAL TRIAL: NCT03184233
Title: Rapid Ventricular Pacing During Cerebral Aneurysm Surgery: a Study Concerning the Safety for Heart and Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Data manager, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/16/205
Record Dates: First submitted 2017-06-02; First posted 2017-06-12 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Pacing, Artificial; Aneurysm, Brain; Arteriovenous Malformations, Cerebral
MeSH Terms: conditions — Intracranial Aneurysm; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: Patients undergoing elective cerebral aneurysm clipping surgery or arteriovenous malformation surgery will be asked to take part and give informed consent.
  A control group of patients undergoing craniotomy without the use of RVP will be built in, having the same exclusion criteria. Both study groups receive a Magnetic Resonance Imaging of the brain pre-and postoperatively as standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebral aneurysm surgery with RVP (Other): Subjects receive a Magnetic Resonance Imaging of the brain pre-and postoperatively as standard of care. To screen for rapid ventricular pacing induced micro-infarcts, the contralateral hemisphere (contralateral to the hemisphere operated on) and fossa posterior will be evaluated. Troponin levels will be determinated preoperatively, peroperative and at 6, 12 and 24 hours postoperative by blood sample. Maximum cTnl level and cTnl level 24 hours will be compared. Brain oxygenation (Sct O₂) by near-infrared spectroscopy will be monitored. During surgery subjects allocated in this study arm will undergo RVP.
  Interventions: Procedure: Rapid ventricular pacing
- Craniotomy without RVP (Active Comparator): Subjects receive a Magnetic Resonance Imaging of the brain pre-and postoperatively as standard of care. To screen for rapid ventricular pacing induced micro-infarcts, the contralateral hemisphere (contralateral to the hemisphere operated on) and fossa posterior will be evaluated. Troponin levels will be determinated preoperatively, peroperative and at 6, 12 and 24 hours postoperative by blood sample. Maximum cTnl level and cTnl level 24 hours will be compared. Brain oxygenation (Sct O₂) by near-infrared spectroscopy will be monitored.
  No rapid ventricular pacing is applied perioperatively.
  Interventions: Procedure: No rapid ventricular pacing

INTERVENTIONS:
Procedure: Rapid ventricular pacing — Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short periods of time during dissection or rupture of the aneurysm. RVP results in an adequate fall in blood pressure which presents as an on-off phenomenon. The technique facilitates the dissection and manipulation of cerebral aneurysms and arteriovenous malformations (AVMs) and can be lifesaving in the case of an intraoperative bleeding or rupture
  Arms: Cerebral aneurysm surgery with RVP
Procedure: No rapid ventricular pacing — No rapid ventricular pacing is applied perioperatively.
  Arms: Craniotomy without RVP

SUMMARY:
Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short periods of time during dissection or rupture of the aneurysm. RVP results in an adequate fall in blood pressure which presents as an on-off phenomenon. However it is not clear whether repetitive periods of pacing are harmless for the patient. Silent cardiac and cerebral infarcts may be undetected. The investigators will study the safety of RVP, particularly for the heart and the brain.

DETAILED DESCRIPTION:
Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short periods of time during dissection or rupture of the aneurysm. RVP results in an adequate fall in blood pressure which presents as an on-off phenomenon. The technique facilitates the dissection and manipulation of cerebral aneurysms and arteriovenous malformations (AVMs) and can be lifesaving in the case of an intraoperative bleeding or rupture. In a former study blood pressure and clinical outcome were used as study parameters. However it is not clear whether repetitive periods of pacing are harmless for the patient. Silent cardiac and cerebral infarcts may be undetected if only clinical outcome is taken as a study parameter. The investigators will study the safety of RVP, particularly for the heart and the brain, using magnetic resonance imaging, brain oxygenation (Sct O₂) evaluated by near-infrared spectroscopy and troponin levels. The purpose of this study is to evaluate the effect of repetitive periods of RVP on the oxygenation of the heart and brain using magnetic resonance imaging, Sct O2 (3) and troponin levels (4) both markers for ischemia damage.

ELIGIBILITY:
Inclusion Criteria:

* elective cerebral aneurysm clipping surgery
* arteriovenous malformation surgery
* craniotomy
* American Society of Anesthesiologists 1,2 and 3

Exclusion Criteria:

* cardiac abnormalities
* coronary heart disease
* valvular heart disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Near infrared spectroscopy | During surgery
  Near infrared spectroscopy measures brain oxygenation (Sct O2), a decrease of more than 10% of the initial Sct O2 or lower than 60% during pacing will be considered as a possible risk of cerebral ischaemia.
Change of cardiac specific enzyme Troponin (cTnl) from preoperative sample(baseline) | A first blood sample is collected immediately preoperative in the operating room. Postoperative samples are taken at 6,12 and 24 hours after start surgery.
  For detection of myocardial injury, the cardiac specific enzyme Troponin (cTnl) is evaluated pre-and postoperatively.

SECONDARY OUTCOMES:
Magnetic resonance imaging | Preoperative and within 1 week post surgery
  Magnetic Resonance Imaging of the brain pre-and postoperatively is used as standard of care. To screen for RVP induced micro-infarcts, the contralateral hemisphere (contralateral to the hemisphere operated on) and fossa posterior will be evaluated.
Occurence of arrhythmias | During surgery
  Any disturbances of the normal rhythmic beating of the heart or myocardial contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp; Tomas Menovsky, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided